CLINICAL TRIAL: NCT05306964
Title: REstrictive Versus LIberal Rate of Extracorporeal Volume Removal Evaluation in Acute Kidney Injury
Acronym: RELIEVE-AKI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was terminated due to insufficient funds.
Sponsor: University of Pittsburgh (Other)
Collaborators: Mayo Clinic (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Raghavan Murugan, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21080010; 1R01DK128100-01A1 (NIH)
Record Dates: First submitted 2022-03-02; First posted 2022-04-01 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Acute Kidney Injury; Fluid Overload; Hypotension; Dialysis; Complications; Critical Illness
Keywords: Fluid overload; Acute kidney injury; Net ultrafiltration; Intensive care unit; Intradialytic hypotension; Complications; Feasibility Trial; Cardiac arrhythmias; Mortality; Dialysis dependence
MeSH Terms: conditions — Acute Kidney Injury; Edema; Hypotension; Critical Illness; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Prospective, two-center, unblinded, parallel-group, 2-arm, comparative effectiveness, stepped-wedge cluster-randomized trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restrictive UFnet Strategy (Active Comparator): Fluid removal will be titrated to keep net ultrafiltration rate between 0.5-1.5 mL/kg/h
  Interventions: Procedure: Restrictive UFnet Rate Strategy
- Liberal UFnet Strategy (Active Comparator): Fluid removal will be titrated to keep net ultrafiltration rate between 2.0-5.0 mL/kg/h
  Interventions: Procedure: Liberal UFnet Rate Strategy

INTERVENTIONS:
Procedure: Restrictive UFnet Rate Strategy — In the restrictive group, the UFnet rate will be titrated between 0.5-1.5 mL/kg/h and maintained throughout fluid removal.
  Arms: Restrictive UFnet Strategy
Procedure: Liberal UFnet Rate Strategy — In the liberal group, the UFnet rate will be titrated between 2.0-5.0 mL/kg/h and maintained throughout fluid removal.
  Arms: Liberal UFnet Strategy

SUMMARY:
Critically ill patients with acute kidney injury and fluid overload who are frequently treated by fluid removal during dialysis are at an increased risk of complications and death. Both slower and faster rates of fluid removal may cause injury to the vital organs. This proposed clinical trial will examine the feasibility of restrictive compared with a liberal rate of fluid removal in order to develop effective treatments for fluid overload and to improve the health of critically ill patients.

DETAILED DESCRIPTION:
"Net ultrafiltration (UFnet)," also known as net fluid removal during kidney replacement therapy, has been used in the treatment of fluid overload among critically ill patients with acute kidney injury (AKI) for more than seven decades. However, the optimal rate of fluid removal (i.e., UFnet rate) remains uncertain, complications such as hypotension and cardiac arrhythmias occur frequently, and more than 40% of patients die. Observational studies in critically ill patients receiving continuous kidney replacement therapy (CKRT) show that UFnet rate has a "J" shaped association with mortality with both slower and faster UFnet rates associated with increased risk of death compared with moderate UFnet rates.

The overall objective of this randomized trial is to establish the feasibility of maintaining patients in the restrictive UFnet rate strategy during treatment with CKRT. The investigator's central hypothesis is that a restrictive UFnet rate strategy embracing a "slow and steady" approach to fluid removal is associated with fewer complications, including cardiac arrhythmias, hypotension, and death, compared with a more liberal "sprint and pause" strategy among critically ill patients.

The trial is a prospective, two-center, unblinded, parallel-group, 2-arm, comparative effectiveness, stepped-wedge cluster-randomized trial among 112 critically ill patients with AKI treated with CKRT in 10 ICUs across two hospital systems. The trial will be conducted at 5 ICUs at University of Pittsburgh Medical Center in Pittsburgh, Pennsylvania, as well as 5 ICUs at Mayo Clinic, Rochester, Minnesota. ICUs will be randomized 1:1 to either a restrictive or a liberal UFnet rate strategy. During the first six months, all ICUs will continue with a liberal UFnet rate strategy. Every two months thereafter or when 10 patients have been enrolled, whichever occurs first, one ICU will be randomized to deploy the restrictive UFnet rate strategy.

In the liberal group, the UFnet rate will be titrated between 2.0-5.0 mL/kg/h and maintained throughout fluid removal. In the restrictive group, the UFnet rate will be titrated between 0.5-1.5 mL/kg/h and maintained throughout fluid removal. The UFnet rates used in both strategies are used in current clinical practice.This feasibility trial will be used to support the rationale and design of a future multicenter phase III randomized trial to examine the effects of alternative UFnet rate strategies on patient-centered clinical outcomes.

Amendment changes- The "Delivered UFnet rates" outcome measure was amended based on a new calculation of effect size when we lowered the sample size from 144 patients to 112 patients in the trial.

The Participant Recruitment Rate Over 21 Months" outcome measure was based on a new sample size estimation when we lowered the sample size from 144 patients to 112 patients in the trial due to slow rate of enrollment in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Stage 3 acute kidney injury according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria
3. Started or intending to start CKRT for volume management
4. Attending intensivist or nephrologist intending to remove net fluid using CKRT for at least 48 hours

Exclusion Criteria:

1. Respiratory distress due to pulmonary edema or fluid overload in unintubated patients
2. Massive volume infusion (i.e., >200 mL/h for >6 hours of continuous infusion)
3. No intention to remove net fluid as determined by attending intensivist or nephrologist
4. Attending intensivist or nephrologist believes that the protocol will not be followed
5. Continuous net fluid removal for >48 hours prior to study enrollment
6. Patients on chronic outpatient hemodialysis
7. Patients with history of, or current admission for kidney transplantation
8. Patients on comfort measures only orders.
9. Moribund not expected to survive >24 hours
10. Confirmed pregnancy
11. Patients treated with extracorporeal membrane oxygenation, ventricular assist device, or intra-aortic balloon pump
12. Organ donors with neurological determination of death (i.e., brain dead donors)
13. Drug overdose requiring CKRT for drug clearance
14. Enrollment in a concurrent interventional clinical trial with direct impact on fluid balance (e.g., >500 mL study drug administration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raghavan Murugan, MD, MS, FRCP, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The RELIEVE-AKI study investigators will review the request for data from other investigators. The investigators will execute a data-sharing agreement with the University of Pittsburgh to share de-identified data with other investigators for research purposes only. The data-sharing agreement will ensure: i.) a commitment to using the data only for research purposes and not to identify any individual participant; ii.) a commitment to securing the data using appropriate computer technology; and iii.) a commitment to destroying or returning the data after analyses are completed on a specific date. The investigators will not release any patient identifiers in any of the data files shared with other researchers. The investigators will also require appropriate confidentiality agreements and approvals from the Institutional Review Boards of other investigators before the data are shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 9 months and ending 36 months after the publication of the primary trial manuscript.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Background] Murugan R, Kerti SJ, Chang CH, Gallagher M, Clermont G, Palevsky PM, Kellum JA, Bellomo R. Association of Net Ultrafiltration Rate With Mortality Among Critically Ill Adults With Acute Kidney Injury Receiving Continuous Venovenous Hemodiafiltration: A Secondary Analysis of the Randomized Evaluation of Normal vs Augmented Level (RENAL) of Renal Replacement Therapy Trial. JAMA Netw Open. 2019 Jun 5;2(6):e195418. doi: 10.1001/jamanetworkopen.2019.5418. PMID 31173127
- [Background] Murugan R, Balakumar V, Kerti SJ, Priyanka P, Chang CH, Clermont G, Bellomo R, Palevsky PM, Kellum JA. Net ultrafiltration intensity and mortality in critically ill patients with fluid overload. Crit Care. 2018 Sep 24;22(1):223. doi: 10.1186/s13054-018-2163-1. PMID 30244678
- [Background] Serpa Neto A, Naorungroj T, Murugan R, Kellum JA, Gallagher M, Bellomo R. Heterogeneity of Effect of Net Ultrafiltration Rate among Critically Ill Adults Receiving Continuous Renal Replacement Therapy. Blood Purif. 2021;50(3):336-346. doi: 10.1159/000510556. Epub 2020 Oct 7. PMID 33027799
- [Background] Naorungroj T, Neto AS, Zwakman-Hessels L, Yanase F, Eastwood G, Murugan R, Kellum JA, Bellomo R. Early net ultrafiltration rate and mortality in critically ill patients receiving continuous renal replacement therapy. Nephrol Dial Transplant. 2021 May 27;36(6):1112-1119. doi: 10.1093/ndt/gfaa032. PMID 32259841
- [Background] Naorungroj T, Neto AS, Zwakman-Hessels L, Fumitaka Y, Eastwood G, Murugan R, Kellum JA, Bellomo R. Mediators of the Impact of Hourly Net Ultrafiltration Rate on Mortality in Critically Ill Patients Receiving Continuous Renal Replacement Therapy. Crit Care Med. 2020 Oct;48(10):e934-e942. doi: 10.1097/CCM.0000000000004508. PMID 32885938
- [Background] Murugan R, Ostermann M, Peng Z, Kitamura K, Fujitani S, Romagnoli S, Di Lullo L, Srisawat N, Todi S, Ramakrishnan N, Hoste E, Puttarajappa CM, Bagshaw SM, Weisbord S, Palevsky PM, Kellum JA, Bellomo R, Ronco C. Net Ultrafiltration Prescription and Practice Among Critically Ill Patients Receiving Renal Replacement Therapy: A Multinational Survey of Critical Care Practitioners. Crit Care Med. 2020 Feb;48(2):e87-e97. doi: 10.1097/CCM.0000000000004092. PMID 31939807
- [Background] Murugan R, Bellomo R, Palevsky PM, Kellum JA. Ultrafiltration in critically ill patients treated with kidney replacement therapy. Nat Rev Nephrol. 2021 Apr;17(4):262-276. doi: 10.1038/s41581-020-00358-3. Epub 2020 Nov 11. PMID 33177700
- [Background] Lumlertgul N, Murugan R, Seylanova N, McCready P, Ostermann M. Net ultrafiltration prescription survey in Europe. BMC Nephrol. 2020 Dec 1;21(1):522. doi: 10.1186/s12882-020-02184-y. PMID 33256635
- [Background] Chen H, Murugan R. Survey of U.S. Critical Care Practitioners on Net Ultrafiltration Prescription and Practice among Critically Ill Patients Receiving Kidney Replacement Therapy. J Crit Care Med (Targu Mures). 2021 Nov 6;7(4):272-282. doi: 10.2478/jccm-2021-0034. eCollection 2021 Oct. PMID 34934817
- [Background] Tehranian S, Shawwa K, Kashani KB. Net ultrafiltration rate and its impact on mortality in patients with acute kidney injury receiving continuous renal replacement therapy. Clin Kidney J. 2019 Dec 17;14(2):564-569. doi: 10.1093/ckj/sfz179. eCollection 2021 Feb. PMID 33623680
- [Background] Naorungroj T, Serpa Neto A, Murugan R, Kellum JA, Bellomo R. Continuous Renal Replacement Therapy: The Interaction between Fluid Balance and Net Ultrafiltration. Am J Respir Crit Care Med. 2021 May 1;203(9):1199-1201. doi: 10.1164/rccm.202011-4097LE. No abstract available. PMID 33513318
- [Background] Kitamura K, Hayashi K, Fujitani S, Murugan R, Suzuki T. Ultrafiltration in Japanese critically ill patients with acute kidney injury on renal replacement therapy. J Intensive Care. 2021 Dec 20;9(1):77. doi: 10.1186/s40560-021-00590-4. PMID 34930481
- [Derived] Murugan R, Chang CH, Raza M, Nikravangolsefid N, Huang DT, Palevsky PM, Kashani K; (RELIEVE-AKI) Study Investigators. Restrictive versus Liberal Rate of Extracorporeal Volume Removal Evaluation in Acute Kidney Injury (RELIEVE-AKI): a pilot clinical trial protocol. BMJ Open. 2023 Jul 7;13(7):e075960. doi: 10.1136/bmjopen-2023-075960. PMID 37419639

RESULTS

PARTICIPANT FLOW:
Recruitment Details: RELIEVE AKI is a multicenter, prospective randomized controlled trial. This study enrolled 99 patients into the study between July 5, 2022 - June 17, 2024 at UPMC and Mayo Clinic hospitals.
Pre-assignment Details: For this study, time of signing the informed consent will be the study enrollment time. There is no patient-level randomization in this trial. The randomization is at the ICU-level and based on study period of every two months.
Groups:
- Sequence 1 (ICU-1): 22 months of Liberal UFnet strategy followed by 1 month of Restrictive UFnet strategy.
- Sequence 2 (ICU-2): 20 months of Liberal UFnet strategy followed by 3 months of Restrictive UFnet strategy.
- Sequence 3 (ICU-3): 14 months of Liberal UFnet strategy and 9 months of Restrictive UFnet strategy.
- Sequence 4 (ICU-4): 8 months of Liberal UFnet strategy and 15 months of Restrictive UFnet strategy.
- Sequence 5 (ICU-5): 23 months of Liberal UFnet strategy and 0 months of Restrictive UFnet strategy.
- Sequence 6 (ICU-6): 12 months of Liberal UFnet strategy and 11 months of Restrictive UFnet strategy.
- Sequence 7 (ICU-7): 18 months of Liberal UFnet strategy and 5 months of Restrictive UFnet strategy.
- Sequence 8 (ICU-8): 6 months of Liberal UFnet strategy and 17 months of Restrictive UFnet strategy.
- Sequence 9 (ICU-9): 10 months of Liberal UFnet strategy and 13 months of Restrictive UFnet strategy.
- Sequence 10 (ICU-10): 16 months of Liberal UFnet strategy and 7 months of Restrictive UFnet strategy.
Period: Step 1: Months 1-6
Arm/Group | Sequence 1 (ICU-1) | Sequence 2 (ICU-2) | Sequence 3 (ICU-3) | Sequence 4 (ICU-4) | Sequence 5 (ICU-5) | Sequence 6 (ICU-6) | Sequence 7 (ICU-7) | Sequence 8 (ICU-8) | Sequence 9 (ICU-9) | Sequence 10 (ICU-10)
Started | 2 | 0 | 2 | 1 | 0 | 1 | 3 | 2 | 0 | 0
Completed | 2 | 0 | 2 | 1 | 0 | 1 | 3 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 2: Months 7-8
Arm/Group | Sequence 1 (ICU-1) | Sequence 2 (ICU-2) | Sequence 3 (ICU-3) | Sequence 4 (ICU-4) | Sequence 5 (ICU-5) | Sequence 6 (ICU-6) | Sequence 7 (ICU-7) | Sequence 8 (ICU-8) | Sequence 9 (ICU-9) | Sequence 10 (ICU-10)
Started | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 (Transition from Liberal to Restrictive UFnet strategy.) | 3 | 0
Completed | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 3: Months 9-10
Arm/Group | Sequence 1 (ICU-1) | Sequence 2 (ICU-2) | Sequence 3 (ICU-3) | Sequence 4 (ICU-4) | Sequence 5 (ICU-5) | Sequence 6 (ICU-6) | Sequence 7 (ICU-7) | Sequence 8 (ICU-8) | Sequence 9 (ICU-9) | Sequence 10 (ICU-10)
Started | 1 | 1 | 0 | 1 (Transition from Liberal to Restrictive UFnet strategy.) | 2 | 4 | 3 | 0 | 1 | 2
Completed | 1 | 1 | 0 | 1 | 2 | 4 | 3 | 0 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 4: Months 11-12
Arm/Group | Sequence 1 (ICU-1) | Sequence 2 (ICU-2) | Sequence 3 (ICU-3) | Sequence 4 (ICU-4) | Sequence 5 (ICU-5) | Sequence 6 (ICU-6) | Sequence 7 (ICU-7) | Sequence 8 (ICU-8) | Sequence 9 (ICU-9) | Sequence 10 (ICU-10)
Started | 3 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 3 (Transition from Liberal to Restrictive UFnet strategy.) | 2
Completed | 3 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 5: Months 13-14
Arm/Group | Sequence 1 (ICU-1) | Sequence 2 (ICU-2) | Sequence 3 (ICU-3) | Sequence 4 (ICU-4) | Sequence 5 (ICU-5) | Sequence 6 (ICU-6) | Sequence 7 (ICU-7) | Sequence 8 (ICU-8) | Sequence 9 (ICU-9) | Sequence 10 (ICU-10)
Started | 2 | 0 | 1 | 0 | 0 | 1 (Transition from Liberal to Restrictive UFnet strategy.) | 3 | 1 | 1 | 0
Completed | 2 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 6: Months 15-16
Arm/Group | Sequence 1 (ICU-1) | Sequence 2 (ICU-2) | Sequence 3 (ICU-3) | Sequence 4 (ICU-4) | Sequence 5 (ICU-5) | Sequence 6 (ICU-6) | Sequence 7 (ICU-7) | Sequence 8 (ICU-8) | Sequence 9 (ICU-9) | Sequence 10 (ICU-10)
Started | 1 | 0 | 1 (Transition from Liberal to Restrictive UFnet strategy.) | 0 | 0 | 3 | 1 | 1 | 1 | 2
Completed | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 7: Months 17-18
Arm/Group | Sequence 1 (ICU-1) | Sequence 2 (ICU-2) | Sequence 3 (ICU-3) | Sequence 4 (ICU-4) | Sequence 5 (ICU-5) | Sequence 6 (ICU-6) | Sequence 7 (ICU-7) | Sequence 8 (ICU-8) | Sequence 9 (ICU-9) | Sequence 10 (ICU-10)
Started | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 0 (Transitioned from Liberal to Restrictive UFnet strategy.)
Completed | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 8: Months 19-20
Arm/Group | Sequence 1 (ICU-1) | Sequence 2 (ICU-2) | Sequence 3 (ICU-3) | Sequence 4 (ICU-4) | Sequence 5 (ICU-5) | Sequence 6 (ICU-6) | Sequence 7 (ICU-7) | Sequence 8 (ICU-8) | Sequence 9 (ICU-9) | Sequence 10 (ICU-10)
Started | 0 | 1 | 0 | 0 | 0 | 0 | 1 (Transition from Liberal to Restrictive UFnet strategy.) | 0 | 5 | 2
Completed | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 9: Months 21- 22
Arm/Group | Sequence 1 (ICU-1) | Sequence 2 (ICU-2) | Sequence 3 (ICU-3) | Sequence 4 (ICU-4) | Sequence 5 (ICU-5) | Sequence 6 (ICU-6) | Sequence 7 (ICU-7) | Sequence 8 (ICU-8) | Sequence 9 (ICU-9) | Sequence 10 (ICU-10)
Started | 1 | 0 (This ICU transitioned from Liberal to Restrictive UFnet strategy.) | 2 | 0 | 0 | 0 | 2 | 0 | 3 | 1
Completed | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Step 10: Month 23
Arm/Group | Sequence 1 (ICU-1) | Sequence 2 (ICU-2) | Sequence 3 (ICU-3) | Sequence 4 (ICU-4) | Sequence 5 (ICU-5) | Sequence 6 (ICU-6) | Sequence 7 (ICU-7) | Sequence 8 (ICU-8) | Sequence 9 (ICU-9) | Sequence 10 (ICU-10)
Started | 1 (This ICU transitioned from Liberal to Restrictive UFnet arm.) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Completed | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of the 99 patients enrolled, the baseline analysis population are the participants who received the intervention (n=95)
Groups:
- Total: Total of all reporting groups
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy | Total
Number analyzed (Participants) | 41 | 54 | 95
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [50 to 71] | 59 [41 to 72] | 59 [46 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 23 | 38
  Male | 26 | 31 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 39 | 50 | 89
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 37 | 49 | 86
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 54 | 95

OUTCOME MEASURES:

1. Primary Outcome: Delivered UFnet Rates.
Description: A minimum separation of 0.53-0.57 mL/kg/h in mean delivered UFnet rates between the two intervention arms.
Time Frame: Until the end of continuous kidney replacement therapy or day 28, whichever occurs first.
Population: The primary outcome was assessed among participants assigned to the Liberal and Restrictive UFnet strategies. Even though the unit of randomization is the ICU, the outcomes were assessed only among participants.
Measure: Median (Inter-Quartile Range); unit: mL/kg/h
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
mL/kg/h | 1.48 [1.00 to 1.94] | 1.57 [0.93 to 2.17]
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.5, GLMM

2. Primary Outcome: No. of Participants With Protocol Deviation.
Description: Protocol deviation defined as delivered UFnet rate that lies >0.5 mL/kg/h outside of the target UFnet rate range for greater than six consecutive hours.
Time Frame: Until the end of continuous kidney replacement therapy or day 28, whichever occurs first.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 4 | 5
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.4, GLMM

3. Primary Outcome: Participant Recruitment/ICU/ 2 Months
Description: An enrollment rate of 1 patient per ICU per time period.
Time Frame: 24 months
Population: Participant recruitment rate per ICU per 2 months during an overall recruitment period lasting 24 months across both treatment arms.
Measure: Mean (Standard Deviation); unit: participant/ ICU/ 2 months
Units Other Than Participants: ICUs
Groups:
- Liberal UFnet Strategy; Restrictive UFnet Strategy: No. of participants recruited per ICU per 2 months
Arm/Group | Liberal UFnet Strategy | Restrictive UFnet Strategy
Number analyzed (Participants) | 56 | 43
Number analyzed (ICUs) | 10 | 9
participant/ ICU/ 2 months | 2.33 (2.11) | 1.79 (1.88)
Statistical Analysis 1: Comparison: Liberal UFnet Strategy; Test type: Other; p = 0.5, GLMM

4. Secondary Outcome: Daily Fluid Balance (Average)
Description: Patient daily fluid balance will be measured while on continuous kidney replacement therapy and reported as average across all study days.
Time Frame: Average daily fluid balance from enrollment to ICU discharge or until day 28, whichever occurs first.
Population: The outcome measure is the average of daily fluid balance (i.e., fluid input minus output over 24 hours) while the patient stayed in the ICU and was compared between the two groups.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
mL | 44 [-1187 to 1202.20] | -53 [-1119.6 to 937.3]
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.3, GLMM

5. Secondary Outcome: Cumulative Fluid Balance
Description: Patient cumulative fluid balance will be measured while on continuous kidney replacement therapy.
Time Frame: Daily from enrollment to ICU discharge or until day 28, whichever occurs first.
Population: This is the cumulative fluid balance (i.e., cumulative fluid input minus output for all days a patient was in the ICU) and was compared between the two groups.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
mL | 229 [-5983 to 7030.8] | 1280.1 [-7390.8 to 6060.4]
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.4, GLMM

6. Secondary Outcome: Duration of Kidney Replacement Therapy
Description: The number of days the patient received kidney replacement therapy while in the hospital.
Time Frame: Daily from enrollment to hospital discharge or until day 28, whichever occurs first.
Population: The secondary outcome was compared among participants assigned to the two groups.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
days | 7 [4 to 17] | 5 [2 to 11]
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.5, GLMM

7. Secondary Outcome: Duration of Mechanical Ventilation
Description: The number of days the patient received mechanical ventilation while in hospital.
Time Frame: Daily from study enrollment to ICU discharge or until day 28, whichever occurs first.
Population: The secondary outcome was compared among participants assigned to the two groups.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
days | 2 [0 to 6] | 3 [0 to 7]
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.3, GLMM

8. Secondary Outcome: Organ Failure Free Days
Description: The no. of days the patient remained free of organ failure while in the ICU.
Time Frame: Daily from study enrollment to ICU discharge or until day 28, whichever occurs first.
Population: The secondary outcome was compared among participants assigned to the two groups.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
days | 3.90 (8.5) | 3.92 (7.9)
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.3, GLMM

9. Secondary Outcome: ICU Length of Stay
Description: The number of days patients need to stay in the ICU
Time Frame: Daily from study enrollment to ICU discharge or day 28, whichever occurs first.
Population: The secondary outcome was compared among participants assigned to the two groups.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
days | 8 [4.5 to 15.5] | 8 [4 to 16]
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.7, GLMM

10. Secondary Outcome: Hospital Length of Stay
Description: The number of days patients need to stay in the hospital
Time Frame: Daily from study enrollment to hospital discharge or day 28.
Population: The secondary outcome was compared among participants assigned to the two groups.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
days | 22.5 [9 to 28] | 16 [5 to 28]
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.2, GLMM

11. Secondary Outcome: Hospital Mortality
Description: The proportion of patients who died while in the hospital.
Time Frame: From study enrollment to hospital discharge or day 28, whichever occurs first.
Population: The secondary outcome was compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 9 | 23
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.02, GLMM

12. Secondary Outcome: Dependence on Kidney Replacement Therapy
Description: The proportion of patients who were on dialysis at hospital discharge.
Time Frame: From study enrollment until hospital discharge or day 28, whichever occurs first.
Population: The secondary outcome was compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 16 | 12
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.2, GLMM

13. Other Pre Specified Outcome: No. of Intradialytic Hypotension Episodes
Description: Intradialytic hypotension will be defined as a new mean arterial pressure <65 mmHg, systolic blood pressure <90 mmHg or a decline in systolic blood pressure >40 mmHg, and/or a >30% increase in dose of existing vasopressors, initiating a new vasopressor, or administration of fluid bolus with a goal to maintain mean arterial pressure >=65 mmHg, systolic blood pressure >=90 mmHg.
Time Frame: From study enrollment until 24 hours after termination of continuous kidney replacement therapy or day 28, whichever occurs first.
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Mean (Standard Deviation); unit: episodes per patient per day
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
episodes per patient per day | 1.16 (0.34) | 1.20 (0.56)
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.7, GLMM

14. Other Pre Specified Outcome: No. of Intradialytic Hypertension Episodes
Description: Intradialytic hypertension will be defined as new onset systolic blood pressure >=160 mmHg or mean arterial pressure >=80 mmHg for more than 1 hour in the absence of any vasopressor or inotrope use.
Time Frame: From study enrollment until 24 hours after termination of continuous kidney replacement therapy or day 28.
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Mean (Standard Deviation); unit: episodes per patient per day
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
episodes per patient per day | 1 (0) | 1.05 (0.32)
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.1, GLMM

15. Other Pre Specified Outcome: No. of Episodes of Intradialytic Cardiac Arrhythmias
Description: New onset intradialytic cardiac arrhythmias including supraventricular tachycardia, bradycardia, atrial fibrillation, ventricular tachycardia, ventricular fibrillation, asystole/pulseless electrical activity will be diagnosed as per American Heart Association.
Time Frame: as for outcome 13
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Mean (Standard Deviation); unit: episodes per patient per day
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
episodes per patient per day | 0.83 (0.29) | 0.92 (0.47)
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.2, GLMM

16. Other Pre Specified Outcome: No. of Participants Who Receive UFnet Rates Higher Than the Assigned Intervention Arm for Treatment of Fluid Overload Emergencies.
Description: No. of participants in whom emergent use of UFnet rates higher than the assigned treatment arm for more than 3 consecutive hours will be noted.
Time Frame: as for outcome 13
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 27 | 8
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p < 0.001, GLMM

17. Other Pre Specified Outcome: No. of Participants With Severe Hypophosphatemia
Description: Hypophosphatemia defined by serum phosphate <0.5 mg/dL
Time Frame: as for outcome 13
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 0 | 0
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0, GLMM

18. Other Pre Specified Outcome: No. of Participants With Severe Hypokalemia
Description: Hypokalemia defined by serum potassium <3.0 mg/dL
Time Frame: as for outcome 13
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 1 | 0
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.5, GLMM

19. Other Pre Specified Outcome: No. of Participants With Severe Hypocalcemia
Description: Hypocalcemia defined by serum calcium <1.90 mg/dL or ionized calcium <0.90 mmol/L
Time Frame: as for outcome 13
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 1 | 1
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.9, GLMM

20. Other Pre Specified Outcome: No. of Episodes of Stopping of CKRT System Due to Hemofilter Clotting or Clogging.
Description: Stopping of CKRT system due to filter clotting and/or clogging.
Time Frame: From study enrollment until termination of continuous kidney replacement therapy or day 28, whichever occurs first.
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Number; unit: Number of episodes
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Number of episodes | 34 | 39
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.8, GLMM

21. Other Pre Specified Outcome: No. of Participants With Discontinuation of Fluid Removal Due to Hemodynamic Instability.
Description: No. of participants in whom fluid removal is stopped due to hemodynamic instability such as intradialytic hypotension, cardiac arrhythmias, or cardiac arrest.
Time Frame: From study enrollment until termination of continuous kidney replacement therapy or day 28, whichever occurs first.
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 21 | 24
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0, GLMM

22. Other Pre Specified Outcome: No. of Participants in Whom Surgical Wounds Are Left Open After Surgery Due to Tissue Edema.
Description: This will be determined as per the primary surgeon. Abdominal wounds left open for a second look or for abdominal re-exploration will not be counted unless there is concurrent tissue edema precluding abdominal closure.
Time Frame: as for outcome 13
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 0 | 0
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0, GLMM

23. Other Pre Specified Outcome: No. of Participants With New Organ Dysfunction as Assessed by Change in Sequential Organ Failure Assessement (SOFA) Scoring System From Baseline.
Description: New organ dysfunction will be assessed by changes in SOFA scores from the baseline across the five organ systems of central nervous system, cardiovascular, respiratory, coagulation, and liver.
Time Frame: as for outcome 13
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 19 | 33
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.2, GLMM

24. Other Pre Specified Outcome: No. of Participants With Worsening of Systolic or Diastolic Cardiac Function on Echocardiogram From Baseline.
Description: Changes in transthoracic echocardiogram will be assessed from baseline (if available)
Time Frame: as for outcome 13
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 0 | 0
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0, GLMM

25. Other Pre Specified Outcome: No. of Participants With Worsening of Pulmonary Edema on Chest X Ray and/or CT Scan Based on Radiologist Report.
Description: Changes in chest X ray and CT scan will be assessed from baseline (if available).
Time Frame: as for outcome 13
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 4 | 6
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.9, GLMM

26. Other Pre Specified Outcome: No. of Participants With Worsening of Ileus on Abdominal X Ray and/or CT Scan Based on Radiologist Report.
Description: Changes in abdominal X ray and CT scan will be assessed from baseline (if available)
Time Frame: as for outcome 13
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 0 | 0
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0, GLMM

27. Other Pre Specified Outcome: No. of Participants With Bowel Ischemia or Anastomotic Breakdown Based on Intraoperative Findings.
Description: Intraoperative findings of bowel ischemia or anastomotic breakdown will be noted as determined by the surgeon (if available).
Time Frame: as for outcome 13
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 1 | 1
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.9, GLMM

28. Other Pre Specified Outcome: No. of Participants With Pressure Ulceration Per Nursing Records.
Description: No. of participants with new diagnosis of pressure ulcerations as documented by the nursing staff in the electronic medical record (if available)
Time Frame: as for outcome 13
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 1 | 0
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0, GLMM

29. Other Pre Specified Outcome: No. of Participants With New Wound Infection Per Nursing Records.
Description: No. of participants with new diagnosis of wound infection as documented by the nursing staff in the electronic medical record (if available)
Time Frame: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 0 | 1
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0, GLMM

30. Other Pre Specified Outcome: No. of Participants With New Arterial and/or Deep Vein Thrombosis as Assessed by Doppler Studies.
Description: New arterial thrombosis or deep vein thrombosis as assessed by doppler study (if available)
Time Frame: as for outcome 13
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 1 | 1
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0, GLMM

31. Other Pre Specified Outcome: No. of Participants With Severe Anemia Requiring Red Cell Transfusions.
Description: Participants with severe anemia requiring red cell transfusions (if available).
Time Frame: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 16 | 26
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.5, GLMM

32. Other Pre Specified Outcome: No. of Participants With Severe Thrombocytopenia Requiring Platelet Transfusions.
Description: No. of participants with severe thrombocytopenia requiring platelet transfusions (if available).
Time Frame: as for outcome 13
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 6 | 15
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.2, GLMM

33. Other Pre Specified Outcome: No. of Participants With New Secondary Infections.
Description: New diagnosis of secondary infections occurring after initiation of study intervention will be collected based on culture data, antibiotic use and suspected sepsis as per clinician judgment (if available).
Time Frame: as for outcome 13
Population: The adverse events were compared among participants assigned to the two groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
Number analyzed (Participants) | 41 | 54
Participants | 3 | 4
Statistical Analysis 1: Comparison: Restrictive UFnet Strategy vs Liberal UFnet Strategy; Test type: Other; p = 0.3, GLMM

ADVERSE EVENTS:
Time Frame: Adverse events for this study were collected from study enrollment until 24 hours after termination of continuous kidney replacement therapy, up to a maximum time frame of 28 days. For example, if continuous kidney replacement therapy was terminated on day 14 on a patient, adverse events were collected until day 15. If continuous kidney replacement therapy continued beyond 28 days, the adverse events were collected only up to 28 days.
Arm/Group | Restrictive UFnet Strategy | Liberal UFnet Strategy
All-Cause Mortality (participants affected / at risk) | 9/43 | 23/56
Serious Adverse Events (participants affected / at risk) | 16/43 | 29/56
Other Adverse Events (participants affected / at risk) | 41/43 | 54/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Restrictive UFnet Strategy (N=43) | Liberal UFnet Strategy (N=56)
Prolonged inpatient hospitalization (General disorders) | 3 | 4
Death after transition to comfort measures (General disorders) | 7 | 13
Subdural hematoma (Vascular disorders) | 2 | 0
End Stage Renal Disease (Renal and urinary disorders) | 0 | 1
Hypoxemic respiratory failure requiring intubation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
New small bowel obstruction (General disorders) | 0 | 1
Cardiopulmonary arrest (Cardiac disorders) | 1 | 2
Multisystem organ failure resulting in death (General disorders) | 2 | 4
Worsening acidosis and hypotension despite up-escalation of pressors (General disorders) | 1 | 0
GI hemorrhage (Gastrointestinal disorders) | 0 | 1
Undifferentiated shock and hypertensive cardiomyopathy (General disorders) | 0 | 1
Hemorrhagic and hypovolemic shock secondary to massive hematemesis from GE varices. (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Restrictive UFnet Strategy (N=43) | Liberal UFnet Strategy (N=56)
Intradialytic hypotension (Cardiac disorders) | 31 | 43
Intradialytic hypertension (Cardiac disorders) | 9 | 16
Cardiac arrhythmias (Cardiac disorders) | 3 | 12
Use of rescue net ultrafiltration (Renal and urinary disorders) | 27 | 8
Severe hypophosphatemia (<0.5 mg/dL) (Metabolism and nutrition disorders) | 0 | 0
Severe hypokalemia (<3.0 mg/dL) (Metabolism and nutrition disorders) | 1 | 0
Severe hypocalcemia (<1.90 mg/dL) (Metabolism and nutrition disorders) | 1 | 1
Hemofilter clotting or clogging (General disorders) | 18 | 21
UFNET discontinuation due to instability (Renal and urinary disorders) | 21 | 24
Surgical wounds edema (Injury, poisoning and procedural complications) | 0 | 0
New organ dysfunction (General disorders) | 19 | 33
Worsening cardiac function (Cardiac disorders) | 0 | 0
Worsening of pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Worsening of ileus (Gastrointestinal disorders) | 0 | 0
Bowel ischemia or anastomotic breakdown (Gastrointestinal disorders) | 1 | 1
New pressure ulcerations (Skin and subcutaneous tissue disorders) | 1 | 0
New wound infections (Skin and subcutaneous tissue disorders) | 0 | 1
New arterial thrombosis (Vascular disorders) | 1 | 0
New venous thrombosis (Vascular disorders) | 0 | 1
Severe anemia (Blood and lymphatic system disorders) | 16 | 26
Severe thrombocytopenia (Blood and lymphatic system disorders) | 6 | 15
New secondary infections (Infections and infestations) | 3 | 4

LIMITATIONS AND CAVEATS:
First, clinicians may hold firm beliefs about UFnet titration, and their awareness of treatment assignment may have led to bias in UFnet titration, specifically not to increase UFnet rates in the liberal arm. Second, we did not assess circulating intravascular volume in UFnet titration as no technology has been validated for net fluid removal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT05306964/Prot_001.pdf
  • Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT05306964/SAP_002.pdf
  • Informed Consent Form (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT05306964/ICF_000.pdf